CLINICAL TRIAL: NCT01118208
Title: Blister Packaging Medication to Increase Treatment Adherence and Clinical Response: Impact on Suicide-Related Morbidity and Mortality
Brief Title: Blister Packaging Medication to Increase Treatment Adherence and Clinical Response
Acronym: BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Peter M. Gutierrez, Clinical/Research Psychologist, VA Eastern Colorado Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: W81XWH-09-1-0723
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Medication Adherence; Accidental Overdose; Deliberate Overdose; Suicide, Attempted
Keywords: Medication adherence; Accidental overdose; Deliberate overdose; Suicide, attempted
MeSH Terms: conditions — Medication Adherence; Suicide, Attempted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blister Packaging (Experimental): Patients will receive all prescription medications on blister pack cards.
  Interventions: Other: Blister packaging medications
- Dispense as Usual (Active Comparator): Patients will receive all prescription medications in standard pill bottles.
  Interventions: Other: Dispense as usual

INTERVENTIONS:
Other: Blister packaging medications — Dispensing prescription medications on pre-filled blister package cards.
  Other Names: Blister cards, bubble packs, unit-dose packaging.
  Arms: Blister Packaging
Other: Dispense as usual — Dispensing prescription medications in standard pill bottles.
  Arms: Dispense as Usual

SUMMARY:
This quantitative, interview-based study will determine if increased prescription medication adherence via blister pack administration will reduce suicide related behavior among the high risk population of patients discharged from a psychiatric inpatient unit. The aims of the project are to determine whether blister packaging medication significantly increases treatment adherence and if blister packaging significantly decreases intentional self-poisoning behavior (i.e., suicide attempts and completions). By tracking former psychiatric inpatients for 12 months post-discharge and obtaining monthly medication adherence ratings, we will determine if blister packaging (BP) medications leads to better adherence than dispensing as usual (DUA). The psychiatric patients we will be recruiting have been diagnosed with, major affective disorder, bipolar affective disorder, post-traumatic stress disorder, or schizophrenia (or any combination of these diagnoses). By tracking former psychiatric patients for 12 months post-discharge and obtaining monthly reports (self-report and medical record review) of suicide-related behaviors, we will determine if patients in the BP condition have less intentional self-poisoning behavior than those in the DAU condition.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* diagnosed with major affective disorder,
* bipolar affective disorder,
* post-traumatic stress disorder, or
* schizophrenia (or any combination of these diagnoses)
* under voluntary status at some point during admission
* currently prescribed medications
* deemed capable of managing their own medications after discharge
* not currently active duty in any branch of the military
* able to correctly answer questions verifying they understand the consent form
* English-Speaking

Exclusion Criteria:

* Under the age of 18
* Not under voluntary status at some point during admission
* Not currently prescribed medications
* Not able to manage their own medications after discharge
* Non-English-speaking
* Currently active duty in any branch of the military
* Inability to correctly answer questions indicating comprehension of information on the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2009-09; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Medication Adherence as assessed with the Brief Adherence Rating Scale (BARS) | monthly for 12 months

SECONDARY OUTCOMES:
Medication overdoses as measured by the Self-Harm Behavior Questionnaire (SHBQ) | monthly for 12 months
  Both accidental and intentional overdoses will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Gutierrez, Ph.D., Principal Investigator — VA VISN 19 MIRECC
Locations (1):
- Denver VA Medical Center, Denver, Colorado, United States

REFERENCES:
- [Result] Gutierrez PM, Wortzel HS, Forster JE, Leitner RA, Hostetter TA, Brenner LA. Blister Packaging Medication Increases Treatment Adherence in Psychiatric Patients. J Psychiatr Pract. 2017 Sep;23(5):320-327. doi: 10.1097/PRA.0000000000000252. PMID 28961661